CLINICAL TRIAL: NCT02566382
Title: Arthrodesis Gleno Humeral Under Arthroscopy in the Sequelae of Plexus Brachial Evaluation of the Technical Feasibility
Brief Title: Preliminary Study of Feasibility of Arthrodesis Scapula-humeral Under Arthroscopy
Acronym: DESEP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufisciency of recruitment
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RB 12.172 DESEP
Record Dates: First submitted 2015-09-29; First posted 2015-10-02 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Arthroscopy Arthrodesis Gleno-humeral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- shoulder arthroscopy arthrodesis (Experimental): The shoulder surgery will be realized under arthroscopy only.
  Interventions: Procedure: arthroscopy arthrodesis of the shoulder

INTERVENTIONS:
Procedure: arthroscopy arthrodesis of the shoulder — The shoulder surgery will be realized under arthroscopy only

SUMMARY:
Arthrodesis shoulder blade/humerus under arthroscopy. Implementation of an external fixative spray at the proximal level in the thorn of the scapula and distal in the diaphysis humerus.

DETAILED DESCRIPTION:
This trial is about the arthrodesis shoulder blade/humerus under arthroscopy. The main aim of this study is to be able to carry out a fusion scapula-humeral supplements in 6 months. It is required to provide the benefice risk over to reduce the hospitalisation 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Patient having a deficit scapula-humeral mobility
* Impossibility of being operated for a preserving nervous surgery
* Patient affiliation with a social security
* Patient who signed inform consent

Exclusion Criteria:

* Patient with No mobility in all the articulations of the shoulder
* Callus malunion of the higher end of the humerus or the glen of the scapula
* Unable to sign an inform consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Radiological fusion gleno humeral on side and front view after the 6th month of the arthroscopy interventional | 6 months
  This outcome will be considered like a success if the investigators get a continuous bone matrix between the humeral head and glenoid on the scapula and bone frame continues between the humeral head and the acromion. This evaluation will be done by radiographies.

SECONDARY OUTCOMES:
Blood loss | 3 days
  The blood loss during and after the surgery will be calculated and will be considered like a success if the total blood loss are less than 600ml.

CONTACTS AND LOCATIONS:
Locations (1):
- Brest university hospital, Brest, Brittany Region, France